CLINICAL TRIAL: NCT03156192
Title: Music Use and Perceived Psycho-social Benefits of Music of Caregivers of Patients in an Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: 4-2016-1028
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Caregivers of ICU Patients
Keywords: Caregivers; Family-centered care; Music use; Psycho-social benefits of music
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers of ICU patients (Experimental): Caregivers (family member) aged over 20 who provides care to ICU patients
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Survey on the level of depression, quality of life, current and past music experiences, and perceived benefits of music in relation to psycho-social needs

SUMMARY:
The purpose of this study is to investigate how family caregivers of ICU patients perceive their psycho-social needs and quality of life, how they use music in their everyday life and perceive music as beneficial to themselves. Participants are adult family members of critically ill patients in ICU. After obtaining the informed consent form, a questionnaire will be distributed to each participant.

DETAILED DESCRIPTION:
The purpose of this study is to investigate how family caregivers of ICU patients perceive their psycho-social needs and quality of life, how they use music in their everyday life and perceive music as beneficial to themselves. Participants are adult family members of critically ill patients in ICU. After obtaining the informed consent form, a questionnaire will be distributed to each participant. The questionnaire consists of Beck Depression Index, Quality of Life scale, and the self-reported items on music use in everyday lives and perceived benefits of music. Based on the completed measures, how caregivers of ICU patients use music and perceive music as beneficial media for their psycho-social health will be analyzed in relation to demographic information and the current level of depression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* primary caregivers (family members) of ICU patients
* aged over 20

Exclusion Criteria:

* the one who have difficulties in verbal communication due to the history of psychiatric illness or cognitive impairment (e.g., dementia)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Index | a single point in time obtaining the questionnaire (1 day)
quality of Life questionnaire | a single point in time obtaining the questionnaire (1 day)
self-reported music use and perceived benefits of music questionnaire | a single point in time obtaining the questionnaire (1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auerbach SM, Kiesler DJ, Wartella J, Rausch S, Ward KR, Ivatury R. Optimism, satisfaction with needs met, interpersonal perceptions of the healthcare team, and emotional distress in patients' family members during critical care hospitalization. Am J Crit Care. 2005 May;14(3):202-10. PMID 15840894
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Davidson JE. Family-centered care: meeting the needs of patients' families and helping families adapt to critical illness. Crit Care Nurse. 2009 Jun;29(3):28-34; quiz 35. doi: 10.4037/ccn2009611. No abstract available. PMID 19487778
- [Background] Chien WT, Chiu YL, Lam LW, Ip WY. Effects of a needs-based education programme for family carers with a relative in an intensive care unit: a quasi-experimental study. Int J Nurs Stud. 2006 Jan;43(1):39-50. doi: 10.1016/j.ijnurstu.2005.01.006. Epub 2005 Sep 22. PMID 16183062